CLINICAL TRIAL: NCT07056738
Title: Longitudinal Characterization of Inner Retina Health in Low Vision Retinitis Pigmentosa Patients to Optimize Retinal Ganglion Cell-based Optogenetic Vision Restoration Therapy
Brief Title: Prospective Exploratory Cohort Study on Ganglion Cell Degeneration in Retinitis Pigmentosa Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Emilie Macé, Professor Dr. Emilie Macé, Department of Ophthalmology, Center of Biostructural Imaging, University Medical Center Goettingen
Other Study IDs: 2025-03803
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; Ganglion cells; Inner retina; Optogenetics
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood serum samples to identify levels of inflammatory markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: imaging — OCT, OCTA, RNFL-OCT, fundus autofluorescence, fundus imaging, flaremeter, fundus and slit lamp examination

SUMMARY:
The aim of this study is an explorative prospective observation of retinal ganglion cell degeneration and/or inner retina degeneration in Retinitis pigmentosa patients. The rate and patterns of progression will be correlated to the outer retina layers as well as clinical and genetic data of patients. Secondary goal is to determine potential parameters for optogenetic treatment eligibility.

ELIGIBILITY:
Inclusion Criteria:

* genetically diagnosed Retintis pigmentosa
* minimum age of 18 years (legal adult age in Germany)
* patient consent for study participation

Exclusion Criteria:

* lack of capacity to consent in participation of study (unconsciousness, mental capacity, mental illness)
* reduced cooperation during imaging or examination
* age under 18 years
* presence of additional retinal diseases
* insufficient imaging quality due to hazy media (cornea, lense)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing Retinitis pigmentosa patients at the University clinic Göttingen. Patients with Retinitis pigmentosa within Pro Retina self-help groups.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Thickness of ganglion cell inner plexiforme layer (GCIPL) in OCT imaging | 6 months intervals, overall time span 5 years
  Measuring the thickness of the ganglion cell inner plexiforme layer (GCIPL) in macula optical coherence tomography (OCT) imaging of the retina.
Thickness of RNFL thickness in OCT imaging | 6 months intervals, overall time span 5 years
  Measuring the thickness of the retinal nerve fiber layer (RNFL) in macular and optic nerve optical coherence tomography (OCT) imaging of the retina.
PD, VD, ICA of the SRP and DRP with OCTA imaging | 6 months intervals, overall time span 5 years
  Perfusion density (PD), vessel density (VD), intercapillary area size (ICA) of superficial retinal plexus (SRP) and deep retinal plexus (DRP) in OCTA imaging (optical coherence tomography angiography)
Thickness and morphology of inner and outer retinal layers measured with OCT, fundus photography, FAF | 6-12 months intervals, overall time span 5 years
  Thickness and morphology of inner and outer retinal layers measured with optical coherence tomography (OCT), fundus photography, fundus autofluorescence (FAF)
Changes in functional parameters such as BCVA | 6 months intervals, overall time span 5 years
  Changes in functional parameters such as best corrected visual acuity
Correlations of outcome 1-5 with clinical data of patients | 6 months intervals, overall time span 5 years
  Find correlations of imaging outcomes with the clinical data of patients, such as sex, age, age of onset of disease
Correlations of outcome 1-5 with genetic data of patients | 6 months intervals, overall time span 5 years
  Find correlations of imaging outcomes with the Retinitis pigmentosa mutation and inheritance pattern of patients
Correlation of outcome 1-5 with inflammatory markers | 6 months intervals, overall time span 5 years
  Correlation of imaging outcomes and disease progression with inflammatory markers collected with serum blood samples and flaremeter as well as slit lamp and fundus examination findings
Correlation of inner and outer retina parameters over time | 6 months intervals, overall time span 5 years
  Correlation of changes in inner retina and outer retina of collected imaging data over time.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Macé, Professor, Principal Investigator — Else Kroener Fresenius Center for Optogenetic Therapies, University Medical Center Goettingen
Locations (1):
- EKFZ Else Kroener Fresenius Center for Optogenetic Therapies, University Medical Center Goettingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No